CLINICAL TRIAL: NCT03859180
Title: A Pilot Study for a Self-Managed Intervention for Anxiety in Parkinson's Disease
Brief Title: Self-Managed Intervention for Anxiety in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HM20014147
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease; Anxiety
Keywords: Anxiety; Self-managed Intervention; Focused Breathing
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Mixed methods, 6 week randomized clinical trial. Using a block size of 4, a computer generated randomization schedule will be generated for an intervention arm and a waitlist arm.
Who Masked: Outcomes Assessor
Masking Description: Assistant performing data checks will mask the random assignments; written on index cards and sealed in security envelope. Opened following informed consent signature obtained and time one outcome measures completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focused breathing intervention group (Experimental): Participants randomized to this group will be taught how to perform focused breathing for the self-management of anxiety and asked to practice for 4 minutes each day during a six week period. They may practice focused breathing in addition to the twice daily practices if they experience anxiety. They will be asked to document in a diary each time they practice focused breathing.
  Interventions: Behavioral: Focused breathing
- Control group (No Intervention): The participants randomized to this group with not be required to perform any additional behaviors for the six week period of the study. After completing post-tests they will be taught how to perform focused breathing for the self-management of anxiety.

INTERVENTIONS:
Behavioral: Focused breathing — Focused breathing is a series of focused, controlled breaths that aid in relaxation. Each participation in this group will be taught how to do focused breathing by the study investigator. Once determined to be able to perform focused breathing, participants will be asked to practice it for 4 minutes, twice a day, for 6 weeks. If they choose to do so, they may practice focused breathing if they become anxious at other times. They will be asked to keep a diary of each time they practice and/or use focused breathing.
  Arms: Focused breathing intervention group

SUMMARY:
A mixed methods randomized controlled feasibility and acceptability study will be conducted to determine the effects of a self-managed, focused breathing intervention on anxiety in persons who have been diagnosed with Parkinson's disease.

DETAILED DESCRIPTION:
This study is being conducted to determine the feasibility and acceptability of using focused breathing as a self managed, non-pharmacologic intervention for anxiety experienced by those with Parkinson's disease. Participants meeting eligibility criteria will be randomized to either an intervention or control group. Those in the intervention group will be taught how to perform focused breathing and asked to practice it twice daily for six weeks for a minimum of four minutes each time. Anxiety, depressive symptoms, sleep, self-efficacy and quality of life with be measured in participants in both the intervention group before beginning to practice focused breathing as well as in the control group. After six weeks of practice the same measurements will be collected from the intervention group. Additionally, intervention participants will participate in a brief interview at the end of their six weeks of practice. Control group participants will be taught how to perform focused breathing six weeks at the end of a six week wait-period, following collection of data using the aforementioned measures..

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* Hoehn & Yahr I, II, & III
* Self report or clinical diagnosis of anxiety
* Ability to speak and read English

Exclusion Criteria:

* Montreal Cognitive Assessment scores less than 26, indicating cognitive impairment
* Persons under the age of 18 are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Parkinson Anxiety Scale (PAS) | 6 weeks following onset of focused breathing twice daily practice.
  This is an 11 question, Likert scale which includes the following responses:
  Not at all or never Very mild or rarely Mild, or sometimes Moderate, or often Severe, or (nearly) always. The tool is has 3 sub-scales designed to measure persistent anxiety, episodic anxiety, and avoidance behavior in Parkinson's disease. It will be administered pre and post intervention for the experimental group and pre and post enrollment for the control group. Scores from 36-48 could indicate the possibility of an anxiety disorder and the need for a clinical evaluation.

SECONDARY OUTCOMES:
Geriatric Depression Scale | 6 weeks
  This is a 25 item, yes/no scale used to measure depressive symptoms. !1 point is scored for each bolded answer (see copy of tool). A score of 0-4 is considered normal; 5-8 suggests mild depressive symptoms; 8-1 moderate depressive symptoms, and 12-15 severe depressive symptoms. Scores of 5 or greater with will be communicated to the patient's Parkinson's provider. It will be administered pre and post intervention for the experimental group and pre and post enrollment for the control group.
Parkinson Sleep Scale - 2 (PSS-2) | 6 weeks
  This is 12 item Likert scale tool used to measure the experience and quality of sleep in individuals with Parkinson's disease. It is a 5 point scale ranging from 0 (very often) to 4 (never). three domains are measured: Motor symptoms at night, Parkinson's disease symptoms at night, and disturbed sleep. Each domain has 5 questions. Range of the domain scores is 0-20; total score range is 0-60. Participants are asked to answer the questions with referral to the past 7 days. Higher scores indicate greater nocturnal disturbance. It will be administered pre and post intervention for the experimental group and pre and post enrollment for the control group.
General Self Efficacy Scale (GSES) | 6 weeks
  This is a 10 question Likert style tool designed to measure self-efficacy, and has the following options:
  Not true at all (1 point) Hardly true (2 points) Moderately true (3 points) Exactly true.(4 points) Responses are made on a 4-point scale; final composite score range from 10 - 40. Higher scores reflect an optimistic self-belief that one can perform a novel or difficult task or cope with adversity. It will be administered pre and post intervention for the experimental group and pre and post enrollment for the control group.
Parkinson's Quality Scale-8 (PDQ-8) | 6 weeks
  This is an eight item Likert response tool designed to measure quality of life in those with Parkinson's disease and has the following options:
  Never Occasionally Sometimes Often Always or cannot do at all It will be administered pre and post intervention for the experimental group and pre and post enrollment for the control group. Answers of the eight items are summed; a score of 0 (0=never) indicates good health; as the score increases (maximum score is 1000 the higher the score the poorer health).

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lynne Robins, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No